CLINICAL TRIAL: NCT05528614
Title: Evaluation of the Results of Simultaneous Pancreatic and Hepatic Resections for Metastatic Neuroendocrine Tumors
Acronym: ReSiPaTNE
Status: Completed | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 8511
Record Dates: First submitted 2022-08-29; First posted 2022-09-06 (Actual); Last update posted 2023-11-08 (Actual); Status verified 2022-08

CONDITIONS: Tumor of Pancreas
Keywords: Tumor of Pancreas; Metastatic neuroendocrine tumors; Hepatic resection; Pancreatic resection
MeSH Terms: conditions — Pancreatic Neoplasms; Neuroendocrine Tumors

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The indications for synchronous liver resection for metastatic neuroendocrine tumors of pancreatic origin remain debated and poorly described in the literature.

The reported mortality of this type of simultaneous resection remains very high, especially when a cephalic duodenopancreatectomy is associated with a hepatic resection (up to 40%). The benefit in terms of survival remains to be evaluated. The ReSiPaTNE study proposes to create a retrospective cohort of simultaneous pancreatic and hepatic resections for metastatic neuroendocrine tumors in order to evaluate the short and long term results of this type of resection. The evaluation of the results of this type of resection may be useful for the selection of patients for treatment.

ELIGIBILITY:
Inclusion criteria:

* Major subjects (≥18 years old)
* Subject having had a first pancreatic resection for NET with resections of synchronous metastases
* Subject having had a first pancreatic resection for NET followed by a delayed resection of synchronous metastases
* Subject who has not expressed his opposition, after being informed, to the reuse of his data for the purposes of this research

Exclusion criteria:

* Subject who expressed their opposition to participating in the study
* Pregnant women
* Subject under safeguard of justice
* Subjects under guardianship or curatorship

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Major subjects (≥18 years old) having had a first pancreatic resection for NET with resections of synchronous metastases
Sampling Method: Non-Probability Sample
Enrollment: 51 (Actual)
Dates: Start 2022-01-13 (Actual); Primary Completion 2022-11-13 (Actual); Study Completion 2023-01-13 (Actual)

PRIMARY OUTCOMES:
Postoperative morbidity and mortality of simultaneous pancreatic and hepatic resectio | Morbidity and mortality at 90 postoperative days

CONTACTS AND LOCATIONS:
Overall Officials: Pietro ADDEO, MD, Principal Investigator — Service de Chirurgie Générale, Hépatique, Endocrinienne et Transplantation - CHU de Strasbourg - France
Locations (1):
- Service de Chirurgie Générale, Hépatique, Endocrinienne et Transplantation - CHU de Strasbourg - France, Strasbourg, France